CLINICAL TRIAL: NCT06307678
Title: EFFECT OF CALCIUM SILICATE-BASED ROOT CANAL MEDICAMENT ON RELEASE OF BONE RESORPTION AND INFLAMMATION MEDIATORS IN PERIAPICAL LESIONS: A RANDOMISED CONTROLLED CLINICAL TRIAL
Brief Title: Effect of Calcium Silicate Based Root Canal Medicament on Inflammatory Mediators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Meltem Sümbüllü, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AtaturkU-DHF-MS-01
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Periapical; Infection
Keywords: intracanal medicament; intracanal dressing; RANKL; osteoprotegerin; TNF alpha; TGF beta; prostaglandin E2
MeSH Terms: conditions — Infections; Camurati-Engelmann Syndrome | interventions — Calcium Hydroxide; calcium silicate

STUDY DESIGN:
Intervention Model Description: two groups: group 1 calcium hydroxide based medicament (control group) group 2: calcium silicate based medicament
Who Masked: Outcomes Assessor
Masking Description: outcome assessments have performed by a investigator who was blinded to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium silicate based medicament (Experimental): Root canal lengths were determined by an electronic apex locator with a 15-K file R25 and R50 Reciproc files were used at working lengths to complete the canal preparation. During instrumentation, the root canals were irrigated with 2 mL 1% NaOCl. To obtain the first samples, 3 sterile paper points were placed into the root canals beyond the 2-mm root apex and were kept in position for 60 seconds. Thereafter, the paper points were cut 4 mm from the tip30.
  Afterward, root canals were dried with paper points, and calcium silicate based medicament was placed in the canals using a file at a distance of 1 or 2 mm less than the root canal length. Next, the coronal cavities were restored with temporary material.
  Seven days later, the medication was mechanically removed using a master apical file. Subsequently, root canals were irrigated.The final samples were collected from the interstitial fluid of the apical tissue as previously described.
  Interventions: Drug: Calcium Silicate
- calcium hydroxide based medicament (Active Comparator): Root canal lengths were determined by an electronic apex locator with a 15-K file R25 and R50 Reciproc files were used at working lengths to complete the canal preparation. During instrumentation, the root canals were irrigated with 2 mL 1% NaOCl. To obtain the first samples, 3 sterile paper points were placed into the root canals beyond the 2-mm root apex and were kept in position for 60 seconds. Thereafter, the paper points were cut 4 mm from the tip30.
  Afterward, root canals were dried with paper points, and calcium hydroxide based medicament was placed in the canals using a file at a distance of 1 or 2 mm less than the root canal length. Next, the coronal cavities were restored with temporary material.
  Seven days later, the medication was mechanically removed using a master apical file. Subsequently, root canals were irrigated.The final samples were collected from the interstitial fluid of the apical tissue as previously described.
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Drug: Calcium Hydroxide — The samples were taken from the interstitial fluid of the apical tissues using 3 paper points before medicament placement.
  Calcium hydroxide based medicament was placed in the canals using a file at a distance of 1 or 2 mm less than the root canal length.
  At the second appointment, medicamentswere removed, and second samplingwas performed using the same method.
  The RANKL/OPG, TNF alpha, TGF beta, PGE2 levels were measured by the enzyme-linked immunosorbent assay, and their ratio was calculated.
  Other Names: calcium hydroxide based medicament group
  Arms: calcium hydroxide based medicament
Drug: Calcium Silicate — The samples were taken from the interstitial fluid of the apical tissues using 3 paper points before medicament placement.
  Calcium silicate based medicament was placed in the canals using a file at a distance of 1 or 2 mm less than the root canal length. At the second appointment, medicaments were removed, and second sampling was performed using the same method.
  The RANKL/OPG, TNF alpha, TGF beta, PGE2 levels were measured by the enzyme-linked immunosorbent assay, and their ratio was calculated.
  Other Names: calcium silicate based medicament group
  Arms: calcium silicate based medicament

SUMMARY:
Calcium hydroxide is generally preferred in endodontics as an intracanal medicament because of its antimicrobial and biological effects. However, the antimicrobial effect of calcium hydroxide is limited.

The aim of this study was to investigate the effects of calcium silicate-based root canal medicament on the release of RANKL/OPG, TNF-α, PGE-2 and TGF-β1 in root canal treated teeth with periapical lesions.

DETAILED DESCRIPTION:
Sixty patients were randomly divided into two groups using a web program according to the medication selected: Calcium silicate based root canal medicament or calcium hydroxide based root canal medicament.

After removing gutta-percha from the root canals, RANKL/OPG, TNF-α, PGE-2 and TGF- β1 samples were taken from the interstitial fluid of the apical tissues using three paper points.

At the second appointment, medicaments were removed and second sampling was performed using the same method. RANKL/OPG, TNF-α, PGE-2 and TGF- β1 levels were measured by enzyme-linked immunosorbent assay and their ratios were calculated.

ELIGIBILITY:
Inclusion Criteria:

Incisor, canine, and premolar teeth that had previously undergone root canal treatment (cases with persistent and secondary disease) and presented with a diagnosis of chronic apical abscess or asymptomatic apical periodontitis were included. Incisor, canine, and premolar teeth with only 1 root canal were included in the study to avoid untreated extra root canals and difficulties in the preparation, obturation, and restoration of molar teeth and to make treatments more standardized.The patients had not used any antibiotics for 3 months before treatment, and patients were obviously free of systemic diseases.

Exclusion Criteria:

Patients were excluded if teeth showed the presence of a root fracture or any swelling, ankyloses, or periodontal pockets deeper than 4 mm. Teeth on which a rubber dam could not be performed were excluded. Patients with allergy to ibuprofen or ciprofloxacin were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
preoperative and postoperative levels of RANKL/OPG ratio | one week
  The amounts of cytokines RANKL and OPG were measured using an enzyme-linked immunosorbent assay kit.
preoperative and postoperative levels of prostaglandinE2 (PGE2) ratio | one week
  The amounts of PGE2 were measured using an enzyme-linked immunosorbent assay kit.
preoperative and postoperative levels of TNF alpha ratio | one week
  The amounts of TNF alpha were measured using an enzyme-linked immunosorbent assay kit.
preoperative and postoperative levels of TGF beta ratio | one week
  The amounts of TGF beta were measured using an enzyme-linked immunosorbent assay kit.

SECONDARY OUTCOMES:
dependent variables (sex, age, teeth number, smoking habit) | one week
  Did the teeth number, age, sex, smoking habit have any effect on pretreatment or posttreatment levels of RANKL/OPG, PGE2, TNF alpha, TGF beta?

CONTACTS AND LOCATIONS:
Overall Officials: meltem sümbüllü, DDS, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Unal O, Sumbullu M, Laloglu E. Effect of tricalcium silicate-based intracanal dressing on bone resorption and inflammatory mediators in periapical lesions: a randomized controlled clinical trial. Odontology. 2025 Oct;113(4):1667-1677. doi: 10.1007/s10266-025-01093-6. Epub 2025 Mar 28. PMID 40155539